CLINICAL TRIAL: NCT00983398
Title: Phase I/II Study of Intra-Arterial Melphalan Given With Intra-Arterial Carboplatin, Osmotic Blood-Brain Barrier Disruption and Delayed Otoprotective Sodium Thiosulfate for Patients With Recurrent or Progressive CNS Embryonal or Germ Cell Tumors
Brief Title: Melphalan, Carboplatin, Mannitol, and Sodium Thiosulfate in Treating Patients With Recurrent or Progressive CNS Embryonal or Germ Cell Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005056; NCI-2013-00790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OHSU-5056; MR00042551; 5056; IRB00005056 (Other: OHSU Knight Cancer Institute); R01NS044687 (NIH)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Central Nervous System Embryonal Neoplasm; Embryonal Tumor With Multilayered Rosettes, C19MC-Altered; Germ Cell Tumor; Medulloblastoma; Medulloepithelioma; Primitive Neuroectodermal Tumor; Recurrent Childhood Central Nervous System Embryonal Neoplasm; Recurrent Malignant Germ Cell Tumor; Recurrent Medulloblastoma; Recurrent Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Neoplasms, Germ Cell and Embryonal; Medulloblastoma | interventions — Carboplatin; Mannitol; Melphalan; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (mannitol, melphalan, carboplatin, STS) (Experimental): Patients receive mannitol IA over 30 seconds, melphalan IA over 10 minutes, and carboplatin IA over 10 minutes. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Treatment repeats every 4-6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Mannitol; Drug: Melphalan; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Carboplatin — Given IA
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Mannitol — Given IA
  Other Names: D-Mannitol; Mannitol, D-; Osmitrol; Resectisol
Drug: Melphalan — Given IA
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sodium Thiosulfate — Given IV
  Other Names: Cyanide Antidote Package; Disodium Thiosulfate; S-Hydril; Sodium Hyposulfate; Sodium Thiosulfate Pentahydrate; Sodium Thiosulphate; Sodothiol; Thiosulfate, Sodium, Pentahydrate; Thiosulfuric Acid Disodium Salt

SUMMARY:
This phase I/II trial studies the side effects and best dose of melphalan when given together with carboplatin, mannitol, and sodium thiosulfate, and to see how well they work in treating patients with central nervous system (CNS) embryonal or germ cell tumors that is growing, spreading, or getting worse (progressive) or has come back (recurrent). Drugs used in chemotherapy, such as melphalan and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Osmotic blood-brain barrier disruption (BBBD) uses mannitol to open the blood vessels around the brain and allow cancer-killing substances to be carried directly to the brain. Sodium thiosulfate may help lessen or prevent hearing loss and toxicities in patients undergoing chemotherapy with carboplatin and BBBD. Giving melphalan together with carboplatin, mannitol, and sodium thiosulfate may be an effective treatment for recurrent or progressive CNS embryonal or germ cell tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of intra-arterial (IA) melphalan given with IA carboplatin, osmotic BBBD and delayed intravenous (IV) sodium thiosulfate (STS) in subjects with recurrent or progressive embryonal and germ cell tumors of the CNS. (Phase I) II. To estimate the response rate in subjects with recurrent or progressive CNS embryonal and germ cell tumors treated with IA carboplatin, IA melphalan, osmotic BBBD and delayed IV STS. (Phase II)

SECONDARY OBJECTIVES:

I. To describe 2-year progression-free survival (PFS) and overall survival (OS) rates in subjects with recurrent or progressive CNS embryonal and germ cell tumors treated with IA carboplatin, IA melphalan, osmotic BBBD and delayed IV STS. (Phase II) II. To describe neuropsychological and audiology outcomes in subjects with recurrent or progressive CNS embryonal and germ cell tumors treated with IA carboplatin, IA melphalan, osmotic BBBD and delayed IV STS. (Phase II) III. To describe the overall toxicity of IA carboplatin and IA melphalan in conjunction with osmotic BBBD and delayed STS chemoprotection in subjects with recurrent or progressive CNS embryonal or germ cell tumors. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of melphalan followed by a phase II study.

Patients receive mannitol IA over 30 seconds, melphalan IA over 10 minutes, and carboplatin IA over 10 minutes. Patients then receive sodium thiosulfate IV over 15 minutes at 4 and 8 hours after carboplatin. Treatment repeats every 4-6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed CNS embryonal tumor (primitive neuroectodermal tumor [PNET], medulloblastoma, atypical teratoid rhabdoid tumor [ATRT], medulloepithelioma, pineoblastoma or ependymoblastoma), or germ cell tumor, are eligible; subjects may be enrolled on study as first-line treatment; diagnosis will be made on the basis of computed tomography (CT)-assisted or stereotactic biopsy, open biopsy, surgical resection, cerebrospinal fluid (CSF) cytology, or elevated tumor markers
* Subjects may be enrolled as part of first-line treatment; those subjects who enroll as first-line treatment will not be restricted from traditional treatments in the future; at least 14 days must have elapsed since completion of cranial radiotherapy and 28 days since completion of chemotherapy; at least 28 days must have elapsed since completion of total spine radiotherapy
* Subjects with no previous radiotherapy treatment must have a consultation with a radiation oncologist or providers must have a discussion in the context of Neuro-Oncology Tumor Board within 60 days prior to start of IA/BBBD chemotherapy to determine the need for radiotherapy prior to or after IA/BBBD
* Glomerular filtration rate (GFR) or creatinine clearance (CrCl) (24 hour urine) greater than 30 ml/min corrected for body surface area
* Absolute granulocyte count >= 1.0 x 10^3/mm^3
* Platelets >= 100 x 10^3/mm^3
* Creatinine < 1.5
* Total bilirubin < 2.0 mg/dl
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 x upper limits of normal
* Subject's Karnofsky performance status (KPS) must be >= 50% (Eastern Cooperative Oncology Group [ECOG] performance score < 3)
* Subjects or their legal guardian must sign a written informed consent in accordance with institutional guidelines
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study treatment and for the duration of study treatment; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* For the phase II portion of the study, subjects must have disease that is evaluable for response; subjects who have had radiation to all sites of disease are not eligible unless there is imaging evidence of active tumor, ie: increased blood volume

Exclusion Criteria:

* Subjects with radiographic signs of excessive intracranial mass effect with associated rapid neurologic deterioration and/or spinal cord block
* Subjects at significant risk with general anesthesia
* Subjects with uncontrolled (over the last 30 days) clinically significant confounding medical conditions
* Subject is pregnant or is lactating
* Subjects who have contraindications to carboplatin, melphalan, or STS

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I) | 6 weeks
  Will be assessed based on the incidence of dose-limiting toxicity, graded using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. All toxicities will be tabulated by event and by overall. The toxicities will also be tabulated by highest grade. The recovery from toxicities (i.e. hematologic toxicities) will also be summarized.
Response rate (Phase II) | Up to 5 years
  Descriptive statistics will be estimated.

SECONDARY OUTCOMES:
Progression free survival rate (Phase II) | Time from first study treatment to evidence of first progression, assessed at 2 years
  Estimation made using Kaplan-Meier product limit estimation. A Cox proportional hazards regression model will be fit to the data to estimate the association of progression free survival and overall survival with baseline demographic and disease characteristics.
Overall survival rate (Phase II) | Time from time of first study treatment until death, assessed at 2 years
  Estimation made using Kaplan-Meier product limit estimation. A Cox proportional hazards regression model will be fit to the data to estimate the association of progression free survival and overall survival with baseline demographic and disease characteristics.
Change in neurocognitive assessment scores (Phase II) | Baseline to 90 days after completion of study treatment
  Quantitative scores, whenever possible, will be derived from each measure and converted to measure-specific Z scores using normative data. Post-treatment Z scores will be subtracted from pre-treatment Z scores to calculate absolute change in neuropsychological test performance. Significant change will be defined as change of 1 standard deviation. These data will be summarized descriptively.
Proportion of patients with ototoxicity (Phase II) | Up to 30 days after completion of study treatment
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Estimated using proportions with associated confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - OHSU Knight Cancer Institute, Portland, Oregon